CLINICAL TRIAL: NCT05536661
Title: Dry Eye and Digital Asthenopia Signs and Symptoms in Gaming Adults. Impact of Tear Substitute Use.
Brief Title: Impact of Tear Substitute Use on Dry Eye in Gamers.
Acronym: HYAGAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Thea, Spain (Industry)
Collaborators: Crossdata (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THEA-HYA-GAMERS-2019-01
Record Dates: First submitted 2022-09-07; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Evaporative Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Preservative free Hyaluronic acid 0.15% artificial tear instilled in both eyes 4 times daily for 3 days
  Interventions: Other: Preservative free hyaluronic acid artificial tear
- Control group (No Intervention): No artificial tear instilation

INTERVENTIONS:
Other: Preservative free hyaluronic acid artificial tear — Ocular lubricant
  Arms: Study group

SUMMARY:
Clinical, prospective, comparative, controlled, single-blind study, on the signs and symptoms of dry eye before and after 3 days of playing video games with the use of artificial tears (Hyabak) versus no intervention.

DETAILED DESCRIPTION:
Adult attendees to a Gamers convention will complete questionnairs and undergo an opthalmological evaluation before and after playing for 3 days in a row. Participants will be randomized into 2 groups of equal size:

1. Study group.
2. Control group. The Study group will instill hyaluronic acid 0.15% artificial tears in both eyes 4 times a day during the 3 days of the video game session, while the control group will not instill artificial tears.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Participants in videogame convention planning to play video games for a minimum of 6 hours daily for the next 3 days.
* Voluntarily accept to participate and sign informed consent form

Exclusion Criteria:

* Ocular, nasolagrimal or palpebral active condition different from dry eye disease.
* History of ocular trauma or infecction in the last 3 months previous to inclusion.
* History of refractive surgery.
* Visual acuity 0.5 or less in at least 1 eye.
* Ocular medication use in the 3 days prior to inclusion.
* History of systemic condition asociated to dry eye.
* Use of systemic medication known to induce dry eye in the last 30 days.
* Known allergy to hyaluronic acid.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
Standard Patient Evaluation of Eye Dryness (SPEED) | Between Day 1 and Day 3
  Change in Standard Patient Evaluation of Eye Dryness (SPEED) score between study and control group (range 0-28, with higher scores indicative of dry eye disease symptoms)

SECONDARY OUTCOMES:
Conjunctival hyperemia measured with McMonnies Chapman scale | Between Day 1 and Day 3
  Change in McMonnies Chapman score (range 0-5, with higher scores indicative of more conjunctival hyperemia) between study and control group
Tear Breakup Time (TBUT) | Between Day 1 and Day 3
  Change in Tear Breakup Time (TBUT) score (normal values > or equal to 10 seconds) between study and control group
Conjunctival staining with lisamine green measured with Oxford scale | Between Day 1 and Day 3
  Change in conjunctival oxford staining score (range 0-5 with higher scores indicative of more staining) between study and control group
Corneal staining with fluorescein measured with Oxford scale | Between Day 1 and Day 3
  Change in corneal oxford staining score (range 0-5 with higher scores indicative of more staining) between study and control group
Schirmer I tear volume test | Between Day 1 and Day 3
  Change in Schirmer score (normal values equal or higher than 10) between study and control group
Near convergence measured with a RAF binocular gauge | Between Day 1 and Day 3
  Change in near convergence between study and control group
Accomodation distance measured with a RAF binocular gauge | Between Day 1 and Day 3
  Change in accomodation distance between study and control group

CONTACTS AND LOCATIONS:
Locations (1):
- Dreamhack Convention, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No